CLINICAL TRIAL: NCT02546791
Title: Frequency and Severity of Pleural Effusion Associated With the Use of Dasatinib in Patients With Chronic Myeloid Leukemia. A Descriptive, Mexican Multicenter Study
Acronym: PASS
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-556
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dasatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic myeloid leukemia patients treated with Dasatinib: patients with a diagnosis of chronic myeloid leukemia treated with Dasatinib for at least 45 days
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
This is a retrospective, multicenter, descriptive analysis of patients with a diagnosis of chronic myeloid leukemia, treated with dasatinib for at least 45 days. The study will include 100 patients treated in different public centers in the Mexican Republic.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥15 years of age
* Diagnosis of chronic myeloid leukemia in any phase that used dasatinib at any time between January 2008 and November 2014
* Have received dasatinib as part of their first-line or second-line treatment for at least 45 days

Exclusion Criteria:

* Patients who received dasatinib as part of any clinical trial
* Patients who do not have complete data on the data collection sheet
* Patients who do not have medical records available at the moment of the data verification

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Public centers in the Mexican Republic
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Detect the absence and presence of pleural effusion in Mexican patients measured from the medical records and databases of each of the participating medical centers | 1 year and 4 month of data collection

SECONDARY OUTCOMES:
Establish the factors associated with response of the patients who develop pleural effusion | 1 year and 4 month of data collection
  Factors:
  Hematological Response
  * Standardization of counts in peripheral blood with leukocytes <10 × 10^9 and platelets <450 ×10^9
  * Absence of immature elements in the smear
  * Basophils <5%
  * Absence of palpable splenomegaly
  Complete Molecular Response (CMR)
  Undetectable BCR-ABL mRNA transcripts by real time quantitative and/or nested Partial Cytogenetic Response (PCR) in two consecutive blood samples of adequate quality (sensitivity >104) Major Molecular Response (MMR)
  Ratio of BCR-ABL to ABL (or other housekeeping genes) ≤0.1% on the international scale
Main characteristics of the patients who develop pleural effusion | 1 year and 4 month of data collection
  Characteristics: Age, gender, comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx